CLINICAL TRIAL: NCT06238648
Title: Multicenter, Randomized Phase II Study of Epcoritamab for Patients With Aggressive B-Cell Lymphomas Achieving a Partial Response After CD19-Directed CAR-T Therapy
Brief Title: Epcoritamab Compared to Observation for Treating B-cell Lymphoma Patients Not in Complete Remission After CD19-directed CAR-T Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-LY-2201; NCI-2023-10170 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-LY-2201 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2024-01-05; First posted 2024-02-02 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Primary Mediastinal Large B-Cell Lymphoma; Transformed Indolent B-Cell Non-Hodgkin Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Watchful Waiting; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (epcoritamab) (Experimental): Patients receive epcoritamab SC on days 1, 8, 15, and 22 of cycles 1-3, days 1 and 15 of cycles 4-9, and day 1 of cycles 10-12. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI at screening, undergo PET/CT and collection of blood samples throughout the trial, and undergo biopsy at screening and end of treatment. Patients may undergo CT or MRI during follow up.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Epcoritamab; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography
- Arm B (observation) (Active Comparator): Patients undergo observation per standard care. Patients also undergo MRI at screening, undergo PET/CT and collection of blood samples throughout the trial, and undergo biopsy at screening and end of treatment. Patients may undergo CT or MRI during follow up.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Patient Observation; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT and/or CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Biological: Epcoritamab — Given SC
  Other Names: Anti-CD20/CD3 Bispecific Antibody GEN3013; DuoBody-CD3xCD20; Epcoritamab-bysp; Epkinly; GEN 3013; GEN-3013; GEN3013
  Arms: Arm A (epcoritamab)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Patient Observation — Undergo observation
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Arm B (observation)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial compares epcoritamab to standard practice (observation) for the treatment of patients with B-cell lymphomas who are not in complete remission after treatment with CD19-directed chimeric antigen receptor T-cell (CAR-T) therapy. Epcoritamab is a bispecific antibody. It works by simultaneously attaching to a molecule called CD20 on cancerous B-cells and a molecule called CD3 on effector T-cells, which are a type of immune cell. When epcoritamab binds to CD20 and CD3, it brings the two cells together and activates the T-cells to kill the cancerous B-cells. Epcoritamab may increase a patient's chances of achieving complete remission after CD19-directed CAR-T therapy, compared to standard observation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare complete response (CR) rate using the Lugano 2014 criteria for patients receiving epcoritamab versus observation alone in patients with aggressive B-cell lymphomas who achieved partial response (PR) post CAR-T therapy.

SECONDARY OBJECTIVES:

I. To compare the progression free survival (PFS) of epcoritamab determined by Lugano 2014 versus observation alone in patients with aggressive B-cell lymphomas post CAR-T.

II. To compare event free survival (EFS) in patients who receive epcoritamab determined by Lugano 2014 versus observation alone in patients with aggressive B-cell lymphomas post CAR-T.

III. To compare the overall survival (OS) of epcoritamab determined by Lugano 2014 versus observation alone in patients with aggressive B-cell lymphomas post CAR-T.

IV. To compare the duration of response (DOR) of epcoritamab determined by Lugano 2014 versus observation alone in patients with aggressive B-cell lymphomas post CAR-T.

V. To compare the duration of complete response (DoCR) of epcoritamab determined by Lugano 2014 versus observation alone in patients with aggressive B-cell lymphomas post CAR-T.

VI. To compare the time to response (TTR) of epcoritamab determined by Lugano 2014 versus observation alone in patients with aggressive B-cell lymphomas post CAR-T.

VII. To compare the objective response rate (ORR) of epcoritamab determined by Lugano 2014 versus observation alone in patients with aggressive B-cell lymphomas post CAR-T.

VIII. To assess the safety and tolerability of epcoritamab post CAR-T in patients with aggressive B-cell lymphomas.

EXPLORATORY OBJECTIVE:

I. To assess outcomes based on CAR-T line of therapy and costimulatory domain of CAR-T construct.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive epcoritamab subcutaneously (SC) on days 1, 8, 15, and 22 of cycles 1-3, days 1 and 15 of cycles 4-9, and day 1 of cycles 10-12. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo magnetic resonance imaging (MRI) at screening, undergo positron emission tomography (PET)/computed tomography (CT) and collection of blood samples throughout the trial, and undergo biopsy at screening and end of treatment. Patients may undergo CT or MRI during follow up.

ARM B: Patients undergo observation per standard care. Patients also undergo MRI at screening, undergo PET/CT and collection of blood samples throughout the trial, and undergo biopsy at screening and end of treatment. Patients may undergo CT or MRI during follow up.

After completion of study treatment, patients are followed up every 90 days for 1 year and then every 180 days for up to 5 years post-registration.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >= 18 years of age
* Documented histological confirmation of diffuse large b-cell lymphoma not otherwise specified [DLBCL NOS], primary mediastinal large b-cell lymphoma (LBCL), or transformations of indolent B-cell lymphomas, according to the 5th edition of World Health Organization (WHO) classification of lymphoid neoplasms, with CD20 positivity as determined by assessment of tumor cells =< 6 months prior to registration pre- CAR-T biopsy specimen by immunohistochemistry or flow cytometry
* Patients treated with the commercially available CD19-directed CAR-T products axicabtagene ciloleucel (axi-cel), tisagenlecleucel (tisa-cel), or lisocabtagene maraleucel (liso-cel), and who have a partial response at day 30 +/- 7 days PET- CT assessment based on Lugano criteria (Deauville score of 4 or 5)
* Documented measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2. (Form is available on the Academic and Community Cancer Research United [ACCRU] web site under Study Resources -> Forms)
* Absolute neutrophil count (ANC) >= 1,000/mm^3, granulocyte colony stimulating factor (G-CSF) allowed (obtained =< 14 days prior to registration)
* Platelet count >= 50,000/mm^3 (obtained =< 14 days prior to registration)
* Hemoglobin >= 7.0 g/dL if asymptomatic or hemoglobin > 8 if symptomatic; transfusion support allowed, if necessary (obtained =< 14 days prior to registration)

  * NOTE: symptoms include shortness of breath, fatigue, lightheadedness
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin or lymphoma involvement of the liver and total bilirubin is =< 5 x ULN (obtained =< 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 x ULN (=< 5 x ULN for patients with liver involvement) (obtained =< 14 days prior to registration)
* Calculated creatinine clearance must be >= 45 mL/min using the Crockcroft- Gault formula (obtained =< 14 days prior to registration)

  * NOTE: If your site laboratory reports use different units of measurement than what is required by the protocol eligibility requirements, please use the "Lab Test Unit Conversion Worksheet" available on the ACCRU website under "General Forms."
* Negative serum pregnancy test done =< 7 days prior to registration for a woman of childbearing potential (WOCBP) only

  * NOTE: A WOCBP is a sexually mature female who:

    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Provide informed written consent =< 28 days prior to registration
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study, i.e., active treatment and clinical follow-up)
* Willing to provide mandatory tissue specimens and blood specimens for correlative research purposes

Exclusion Criteria:

* Patients post CAR-T who have bulky disease defined as a disease focus >= 7.5cm in diameter at day 30 +/- 7 days PET-CT assessment
* Patients post CAR-T who have progressive disease, stable disease or complete response at day 30 +/- 7 days PET-CT assessment based on Lugano criteria
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic, and teratogenic effect on the developing fetus and newborn are unknown

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception (men and women)
* Any of the following prior therapies:

  * CD20xCD3 bispecific antibody at any point prior to registration
  * CD20-targeted monoclonal antibody (e.g., rituximab, obinutuzumab or biosimilars) =< 4 weeks prior to registration
* Ongoing cytokine release syndrome (CRS) or neurotoxicity post CAR-T
* Prior grade 4 CRS or neurotoxicity after most recently administered CAR-T
* Primary central nervous system (CNS) lymphoma or CNS involvement by lymphoma at screening and based on clinical symptoms, MRI, or lumbar puncture
* Co-morbid systemic illness or other severe concurrent disease which, in the judgement of the investigator, would make the patient inappropriate for entry into the study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring systemic treatment (excluding prophylactic treatment) =< 14 days prior to registration, including COVID- 19 infection.

    * NOTE: If evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable and on suppressive therapy.
    * NOTE: If history of treated hepatitis C virus (HCV) infection, HCV viral load must be undetectable.
    * NOTE: Patients known to be human immunodeficiency virus (HIV) positive, but stable on anti-retroviral therapy with an undetectable HIV viral load pre-CART, are eligible for this trial.
    * NOTE: Simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted if responding to active treatment
    * NOTE: Past COVID-19 infection may be a risk factor, but if resolved symptoms and the subject is vaccinated, they may be enrolled
  * Symptomatic congestive heart failure (New York Heart Association [NYHA] class 3 or 4)
  * Unstable angina pectoris
  * Unstable cardiac arrhythmia present =< 14 days prior to registration
  * Psychiatric illness/social situations that would limit compliance with study requirement
  * History or presence of CNS disorder such as seizure disorder (not including resolved childhood febrile seizures), cerebrovascular ischemia/hemorrhage (not including transient ischemic attacks), cerebellar disease, or any autoimmune disease with CNS involvement
* Receiving any other investigational agent which would be considered treatment for the primary neoplasm =< 14 days prior to registration
* Other active malignancy requiring therapy < 2 years prior to registration (localized non-melanoma skin cancer is allowed)
* Clinically significant cardiovascular disease, including: Myocardial infarction within 1 year prior to randomization, or unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association class III-IV) cardiac arrhythmia (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0 grade 2 or higher), or clinically significant electrocardiogram (ECG) abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective status of complete response (CR) | From randomization up to one year
  CR will be assessed using Lugano 2014 criteria. Complete response rate is defined as the number of patients who achieve objective status of CR divided by the total number patients in each arm. Primary analysis population will be used for this endpoint. The proportion of CR rate in each arm with corresponding confidence interval and p-value comparing the CR rate will be reported.

SECONDARY OUTCOMES:
Progression free survival | From randomization to documentation of disease progression or death, assessed up to 5 years post-registration
  Disease progression will be defined by Lugano 2014 criteria. Primary analysis population will be used for this endpoint. The distribution of progression free survival will be estimated using the method of Kaplan-Meier. Progression free survival will be compared between the 2 treatment arms using the log-rank test. The median progression free survival and corresponding 95% confidence intervals will be reported.
Event free survival | From randomization to documentation of disease progression, start of non-protocol lymphoma therapy, or death due to any cause, assessed up to 5 years post-registration
  Disease progression will be defined by Lugano 2014 criteria. Primary analysis population will be used for this endpoint. The distribution of event free survival will be estimated using the method of Kaplan-Meier. Event free survival will be compared between the 2 treatment arms using the log-rank test. The median event free survival and corresponding 95% confidence intervals will be reported.
Overall survival | From randomization to death due to any cause, assessed up to 5 years post-registration
  Primary analysis population will be used for this endpoint. The distribution of overall survival will be estimated using the method of Kaplan-Meier. Overall survival will be compared between the 2 treatment arms using the log-rank test. The median overall survival and corresponding 95% confidence intervals will be reported.
Duration of response | From first documentation of objective status of partial response (PR) or CR to documentation of disease progression, assessed up to 5 years post-registration
  Disease progression will be defined by Lugano 2014 criteria. Primary analysis population achieving response of CR or PR will be used for this endpoint. The distribution of duration of response will be estimated using the method of Kaplan-Meier. Duration of response will be compared between the 2 treatment arms using the log-rank test. The median duration of response and corresponding 95% confidence intervals will be reported.
Duration of complete response | From first documentation of objective status of CR to documentation of disease progression, assessed up to 5 years post-registration
  Disease progression will be defined by Lugano 2014 criteria. Primary analysis population achieving response of CR will be used for this endpoint. The distribution of duration of complete response will be estimated using the method of Kaplan-Meier. Duration of complete response will be compared between the 2 treatment arms using the log-rank test. The median duration of complete response and corresponding 95% confidence intervals will be reported.
Time to response | From randomization to the first documentation of objective status of PR or CR, assessed up to 5 years post-registration
  Response will be defined by Lugano 2014 criteria. Primary analysis population achieving response of CR or PR will be used for this endpoint. The distribution of time to response will be estimated using descriptive statistics such as median and range. Time to response will be compared between the 2 treatment arms using the Wilcoxon-rank sum test.
Objective response rate (ORR) | From randomization up to one year
  Response will be defined by Lugano 2014 criteria. ORR is defined as the number of patients who experience objective response divided by the number of patients in primary analysis population. ORR will be compared between the 2 treatment arms. Confidence intervals for ORR will be calculated according to the approach of Clopper and Pearson. Overall response rate and the corresponding 95% confidence interval will be reported.
Incidence of adverse events | Up to 1 year post-treatment
  Primary analysis population will be used for adverse event analyses. The overall adverse event rates for grade 3 or higher adverse events will be reported. Further analysis of adverse event rates will be considered exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz S Nowakowski, Principal Investigator — Academic and Community Cancer Research United
Locations (6):
- United States (6):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah